CLINICAL TRIAL: NCT04450979
Title: A Randomised, Double-blinded, Parallel Group, Placebo-Controlled Study to Evaluate the Effects of a Bioactive Peptide on Symptoms of Digestive Discomfort in the Elderly
Brief Title: Study to Evaluate Bioactive Peptides' Effect on Digestive Discomfort Symptoms of the Elderly
Acronym: Inflammaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nuritas Ltd (Industry)
Collaborators: Atlantia Food Clinical Trials (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Prevention
Other Study IDs: AFCRO-063
Record Dates: First submitted 2020-06-25; First posted 2020-06-30 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Abdominal Pain
MeSH Terms: conditions — Abdominal Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bioactive hydrolysate (Active Comparator): 20 g of hydrolysed rice protein
  Interventions: Dietary Supplement: Bioactive hydrolysate
- Placebo (Placebo Comparator): 20 g micro crystalline cellulose
  Interventions: Dietary Supplement: Bioactive hydrolysate

INTERVENTIONS:
Dietary Supplement: Bioactive hydrolysate — Participants given a bioactive vegetable hydrolysate to take one dose each morning and one dose each evening for the duration of the study.

SUMMARY:
This trial will investigate the potential of a bioactive peptide to reduce symptoms of digestive discomfort in a generally healthy elderly population. Participants will consume the bioactive peptide for 12 weeks and various measures indicating an improvement in health and well being will be taken throughout the trial. It is believed that consumption of the study product will reduce the severity of digestive discomfort, reduce chronic inflammation, improve blood glucose metabolism and improve physical performance.

DETAILED DESCRIPTION:
Forty subjects aged between 65 and 75 with self-reported symptoms of digestive discomfort will be randomised. Subjects will be randomised to receive either the Bioactive peptide or placebo for a total of 12 weeks.

Subjects will undergo an initial phone screen and will be asked questions regarding their age and their symptoms of digestive discomfort. Eligible subjects will be scheduled for a screening visit. The study will involve 5 visits over a 13 to 16 week period.

At the screening visit (Visit 1) the inclusion and exclusion criteria will be reviewed and the overall details of the study will be explained and informed consent obtained. Vitals and Medical history, demographic data and concomitant medication will be recorded.

Subjects will be asked questions relating to their digestive symptoms, including symptoms of abdominal pain, discomfort, bloating and flatulence. Subjects will complete the Digestive Symptom Frequency Questionnaire (DSFQ), the International Physical Activity Questionnaire (IPAQ) and the Mini-mental State Exam (MMSE) will be administered. The Fried Frailty score will be completed and the Short Physical Performance Battery (SPPB) test will be performed. A fasting blood sample (9mls) will be collected and haematology, biochemistry, glucose and blood lipids will be measured.

Subjects will be provided with a stool collection kit and instructions for collecting and storing. Subjects will collect a stool sample at home, within 24 hours of their next visit and bring it to the clinic at their next visit.

If the subject meets the eligibility criteria, they will be invited to participate in the study and will be given an appointment to return to the study site within 4 weeks for their baseline/week 0 visit.

Subjects will attend visit 2 fasting. The inclusion and exclusion criteria will be reviewed and eligibility for study entry confirmed. An Oral Glucose Tolerance Test will be performed. Haematology, biochemistry and blood lipids will also be measured.

A urine sample will be collected and also stored frozen for analysis of metabolites.

Vitals, anthropometric measurements, concomitant medication and any adverse events will be recorded and The Short Physical Performance Battery (SPPB) test will be performed.

Subjects will complete the Digestive Symptom Frequency Questionnaire and the hand-grip and chair-stand tests will be performed. A DEXA scan will be performed and muscle and fat mass recorded.

Subjects will be randomized to receive the Bioactive peptide or placebo and receive a 4 week supply of product and instructions for dosing. Subjects will be provided with a stool collection kit and instructions for collecting and storing. Subjects will collect a stool sample at home, within 24 hours of their next visit and bring it to the clinic at their next visit.

Subjects will return for visits at week 4, week 8 and week 12.

A similar regimen will be followed for visits at week 4, week 8 and week 12.

The site, investigator, protocol, informed consent form and any other pertinent documents for this study will be approved by: Cork Research Ethics Committee of the Cork Teaching Hospitals, Lancaster Hall, 6 Little Hanover Street, Cork.

The investigator is responsible for ensuring that all source documents (i.e. study and/or medical records) are completed and maintained according to the study protocol, Good Clinical Practice (GCP) and are available at the site.

LIST OF ABBREVIATIONS AND DEFINITION OF TERMS

ANCOVA Analysis of co-variance AUC Area Under the Plasma Concentration BMI Body mass index BP Blood pressure CI Confidence interval CRF Case Report Form CRO Contract Research Organization EFSA European Food Safety Authority GCP Good Clinical Practice GMP Good Manufacturing Practice HbAIc Glycated haemoglobin (A1c) ICH International Conference on Harmonization INCI The International Nomenclature of Cosmetic Ingredients ITT Intent-to-treat kDa Kilodalton kg Kilogram L Liter MCH Mean corpuscular hemoglobin MCHC Mean corpuscular hemoglobin concentration MCV Mean corpuscular volume MCPs Marine collagen peptides MedDRA Medical Dictionary for Regulatory Activities mITT Modified intention-to-treat mL Milliliter mmHg Millimeter of mercury mmol/mol Millimoles per mole OGTT Oral glucose tolerance test PPP Per protocol population RDW Red cell distribution width SAE Serious adverse event SAP Statistical analysis plan VLDL Very low-density lipoprotein WHO World Health Organisation

ELIGIBILITY:
Inclusion Criteria:

* Be able to give written informed consent
* Be between 65 and 75 years of age (inclusive)
* Have symptoms of digestive pain & discomfort
* Have a Fried Frailty score of <2
* Have a Short physical performance battery (SPPB) score of >5 and <10
* Have a Mini Mental State Exam (MMSE) score >24
* Have low or moderate activity according to the IPAQ short form
* Have a BMI <30 kg/m2
* Be in good general health.

Exclusion Criteria:

* Are less than 65 and greater than 75 years of age
* Are severely immunocompromised (HIV positive, transplant Subject, on antirejection medications, on a steroid for >30 days.
* Have a diagnosis of Irritable Bowel Syndrome
* Is taking a high dose of statins and/or has changed had their dose modified in the previous 6 months
* Is experiencing muscle pain, soreness or muscle loss in the previous 6 months
* Has a history of drug and / or alcohol abuse at the time of enrolment
* Has changed their dietary habit within the preceding month
* Has a known organic disease, including an inflammatory bowel disease, a benign or malign tumour of intestine or colon and significant systemic disease
* Subject currently involved in any other clinical trial or having participated in a trial within the preceding 90 days
* Has known allergy to components of the test product
* Use of anti-inflammatory steroid medications, anticoagulants, current/recent (3 months) history of anabolic steroid, corticosteroid or estrogen use, testosterone replacement therapy (ingestion, injection, or transdermal), or any anabolic steroid
* Has any concurrent medical or psychiatric condition that, in the opinion of the Investigator, would compromise his/her ability to comply with the study requirements

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-06-14 (Actual); Primary Completion 2016-10-28 (Actual); Study Completion 2017-01-20 (Actual)

PRIMARY OUTCOMES:
Digestive symptom frequency questionnaire | Baseline (week 0) and end of treatment (week 12)
  The primary endpoint is the difference between the change experienced over 12 weeks in the active group versus the change in the placebo group using the digestive symptom frequency questionnaire (DSFQ) at baseline and end of treatment

SECONDARY OUTCOMES:
To determine the effect of supplementation of a Bioactive Peptide on muscle mass | Baseline (week 0) and week 12
  Muscle mass, measured by dual-energy x-ray absorptiometry (DXA) at weeks 0 and 12
To determine the effect of supplementation of a Bioactive Peptide on upper body muscle strength | Baseline (weeks 0) and week 4, week 8 and week 12
  Upper body muscle strength, measured by the hand-grip test
To determine the effect of supplementation of a Bioactive Peptide on lower body muscle strength | Baseline (weeks 0) and week 4, week 8 and week 12
  Lower body muscle strength, measured by the chair stand test
To determine the effect of supplementation of a Bioactive Peptide on physical performance | Baseline (weeks 0) and week 12
  Short physical performance battery test score
To determine the effect of supplementation of a Bioactive Peptide on blood glucose | Baseline (weeks 0) and week 12
  Glucose as measured by the Oral Glucose Tolerance Test
To determine the effect of supplementation of a Bioactive Peptide on blood markers of inflammation | Baseline (weeks 0) and week 4, week 8 and week 12
  Inflammatory cytokines (IL6 & IL1R, CRP, TNF)
To determine the effect of supplementation of a Bioactive Peptide on blood lipid | Baseline (weeks 0) and week 4, week 8 and week 12
  Lipids (Total cholesterol, LDL, HDL, Triglycerides